CLINICAL TRIAL: NCT05356104
Title: GLP-1 Analogue in Preventing Progression of Small Vessel Disease (GAPP-SVD) - A Pilot Study
Brief Title: GLP-1 Analogue in Preventing Progression of Small Vessel Disease (GAPP-SVD)
Acronym: GAPP-SVD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAPP-SVD
Record Dates: First submitted 2022-04-08; First posted 2022-05-02 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Small Vessel Disease
Keywords: cSVD
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Intervention Model Description: 110 patients with cSVD of Age-Related White Matter Changes Scale of 2 or 3 will be randomized into "treatment arm" with GLP-1R agonist and standard medical therapy, and "control" arm with standard medical therapy alone in a 1:1 ratio. In this 78 weeks pilot study, investigators shall evaluate the tolerability and safety profile of exenatide, a GLP-1R agonist in SVD patients, together with changes in clinical, imaging and sonographic parameters.
Who Masked: Outcomes Assessor
Masking Description: Assessors for TCD and Cognition and behavior assessments will be blinded to the randomization assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exenatide extended release (Active Comparator): Prescribe study drug: Exenatide extended release. The dosage and frequency is 2mg once weekly via subcutaneous injection for 78 weeks
  Interventions: Drug: Exenatide extended release
- Standard of care (No Intervention): Standard medical therapy

INTERVENTIONS:
Drug: Exenatide extended release — 2mg once weekly via subcutaneous injection
  Other Names: Bydureon BCise
  Arms: Exenatide extended release

SUMMARY:
Cerebral small vessel disease (cSVD), a result of neurovascular cell dysfunction, is a major cause of stroke, dementia and mobility problems worldwide. Vascular risk factor control alone may not be sufficient to prevent the development of vascular cognitive impairment (VCI) in patients with cSVD according to previous clinical trials.

The presence of glucagon-like peptide-1 receptor (GLP-1R) in cerebral microglia may reveal a potential therapeutic target for prevention of cSVD progression and its disabling clinical outcomes. At the cellular and animal experimentation levels, GLP-1R agonist demonstrated reversal of some pathogenic processes in cSVD. However, its application to cSVD patients remains to be elucidated.

Investigator aims to investigate the safety and efficacy of GLP-1R agonist in patients with moderate-to-severe cSVD.

DETAILED DESCRIPTION:
In this single-center, open-label (assessor blinded), randomized controlled study, 110 patients with cSVD of Age-Related White Matter Changes Scale of 2 or 3 will be randomized into "treatment arm" with GLP-1R agonist and standard medical therapy, and "control" arm with standard medical therapy alone in a 1:1 ratio. In this 78 weeks pilot study, investigators shall evaluate the tolerability and safety profile of exenatide, a GLP-1R agonist in SVD patients, together with changes in clinical, imaging and sonographic parameters.

Clinical and biochemical measures will be assessed at baseline, 12 weeks, 26 weeks and 52 weeks. Transcranial Doppler Ultrasound (TCD) will be performed at baseline, 12 weeks, 26 weeks, 52 weeks and 78 weeks. MRI will be performed at baseline and 78 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Chinese ethnicity;
2. Age 55 to 80 years old;
3. Age-Related White Matter Change (ARWMC) Scale of 2 or early 3 in FLAIR MRI;
4. Modified Functional Ambulation Classification 5 or above;
5. Montreal Cognitive Assessment (MoCA) score < 25;
6. Both diabetic and non-diabetic patient are eligible;
7. Patient who understands the purpose and requirements of the study, and able to provide an informed consent;

Exclusion Criteria:

1. Dementia or MoCA score lower than 2nd percentile of the age and education adjusted cutoff ;
2. Cerebral white matter changes unrelated to neurodegenerative, e.g. CADASIL, X-linked adrenoleukodystrophy, metabolic diseases, multiple sclerosis, etc.;
3. Contraindication to GLP-1R agonist, including thyroid carcinoma, pancreatic pathology, proliferative retinopathy, hypersensitivity to GLP-1R agonist and history of family history of multiple endocrine neoplasia;
4. BMI <18.5kg/m2;
5. Contraindication to proposed imaging, e.g. chronic kidney disease (KDNIGO) stage 4 or above, acute kidney injury, hypersensitivity to gadolinium-based contrast, non-MRI conditional implants or prosthesis;
6. Medical condition that would not allow the patient to adhere to the protocol or complete the study.;
7. Patient with established neurodegenerative disorders (e.g. Parkinson's Disease, Alzheimer's Disease, etc.);
8. Pregnancy.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of Brain Peak Width of Skeletonized Mean Diffusivity | Baseline and week 78
  Peak Width of Skeletonized Mean Diffusivity is a robust, fully-automated and easy-to-implement marker for cerebral small vessel disease based on diffusion tensor imaging, white matter tract skeletonization and histogram analysis. It is a biomarker for brain MRI images.

SECONDARY OUTCOMES:
Number of recurrent stroke | Baseline and week 78
  Record of any recurrent stroke from medical note/system
Change of Hong Kong MOntreal Cognitive Assessment | Baseline, week 12, week 26, week 52 and week 78
  Hong Kong MOntreal Cognitive Assessment (HK-MoCA) is a cognitive assessment tool. Score from 0 to 30 . The lower score reflect the worse the outcome.
Change The Chinese Geriatric Depression Scale 30 | Baseline, week 12, week 26, week 52 and week 78
  The Chinese Geriatric Depression Scale is used to detect depressive mood. Score 0 to 30. The higher the score, the worse the outcome
Change of Pittsburgh sleep quality index | Baseline, week 12, week 26, week 52 and week 78
  Pittsburgh sleep quality index Chinese Version is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The questionnaire contains frequency questions related to sleep quality, each question scale from 0 to 3. The higher the score, the worse the outcome. There is no total score available for this assessment
Change of Hong Kong List Learning Test | Baseline, week 12, week 26, week 52 and week 78
  Hong Kong List Learning Test s a newly developed Chinese memory test designed for the assessment of the processes and organizational strategies involved in learning verbal information. The more negative the standard deviation the worse the outcome
Change of Neuropsychiatric Inventory | Baseline, week 12, week 26, week 52 and week 78
  Neuropsychiatric Inventory is a brief interview with a family member or friend who knows the study subject . It is used to measure behavioral symptoms. It evaluates 12 behavioral areas commonly affected in patients with dementia. It evaluates the frequency (scale from 1 to 4), severity (scale from 1 to 3), distress to caretaker (scale from 1 to 5) of each behavioral symptom.
  The higher the score of any area means the worse outcome. There is no total score available for this assessment
Change of disability assessment for dementia | Baseline, week 12, week 26, week 52 and week 78
  Disability assessment for dementia evaluates 11 basic daily activities of elderly people with dementia. It evaluates each activity in 3 stages: initiation, planning and organization, effective performance. Score 1 or 0 for each question.
  The higher the total score, the better the outcome. The total score is from 0 to 47.
Change of Gait | Baseline, week 12, week 26, week 52 and week 78
  Gait velocity will be assessed using the 8-meter walking time. Time for walking 8-m will be measured by a stopwatch. The faster of two trials will be used in the analysis
  The faster of the walking time the better outcome.
Change of balance | Baseline, week 12, week 26, week 52 and week 78
  Single leg stance time will be measured by asking individuals, with their hands on their hips, to balance as long as possible on one leg with an upper limit of 30 seconds. Two trials for each leg will be performed. The best time of the four trials will be used for analysis. The longer to time duration the better outcome.
Change of Pulsatility Index | Baseline, week 12, week 26, week 52 and week 78
  Pulsatility Index of Transcranial doppler ultrasound is a painless test that uses sound waves to detect medical problems that affect blood flow in your brain. It is a measure of vascular resistance of cerebral vessels. The higher the index means higher resistance and stiffness of blood vessels which lead to worse outcome. There is no minimum or maximum values available for this index.
Change of Breath Holding Index | Baseline, week 12, week 26, week 52 and week 78
  Breath Holding Index calculated based on the mean flow velocities of the middle cerebral artery using transcranial Doppler. It indicates the brain artery could react better to lowered oxygen level. The higher the index means better reaction to lowered oxygen level which leads to better outcome. There is no minimum or maximum values available for this index.
Change of DNA methylation | Baseline, week 12, week 26, week 52 and week 78
  blood biomarker. DNA methylation-derived epigenetic age clock is an indicator of biological aging.
Change of neurovascular inflammation | Baseline, week 12, week 26, week 52 and week 78
  blood biomarker to investigate neurovascular inflammation that induce neurodegeneration

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Yiu Ming Ip, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No